CLINICAL TRIAL: NCT06757127
Title: Enhancing Surgical Outcomes with a Closed-Loop Audit of ERAS Protocols in Emergency Laparotomy At a Conflict-Affected Hospital
Brief Title: Quality Improvement Audit of ERAS Protocol Adherence in Emergency Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudan Medical Specialization Board (Other Government)
Responsible Party: Principal Investigator, Alsadig Suliman, Principal Investigator, Sudan Medical Specialization Board
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: ALNAO-EC-2024-09; ANH/EC/2024/082 (Other: Alnao Teaching Hospital)
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Emergency Laparotomy; Quality Improvement; Implementation Science; Enhanced Recovery After Surgery (ERAS) Protocol
Keywords: Enhanced Recovery After Surgery (ERAS); Emergency Laparotomy; Resource-Limited Settings; Patient-Centered Care; Audit and Compliance; Surgical Care Optimization
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Intervention Assessment of Staff Adherence to ERAS Protocol in Emergency Laparotomy (Other): This arm involves evaluating the baseline adherence of healthcare staff, including doctors, nurses, and anesthesia technicians, to the ERAS protocols for emergency laparotomy patients. Data collection was exclusively based on direct observation to assess adherence accurately while minimizing any observer effect that might alter staff behavior. A checklist based on ERAS ® Society guidelines for emergency laparotomy, tailored to the resource constraints of the setting, was used to assess compliance with criteria across preoperative, intraoperative, and postoperative phases. No intervention was applied during this phase, serving as a baseline for comparison with post-intervention outcomes
  Interventions: Other: ERAS Protocol Adaptation for Emergency Laparotomy
- Post-Intervention Assessment of Staff Adherence to ERAS Protocol in Emergency Laparotomy (No Intervention): This arm evaluates the adherence of healthcare staff to the ERAS protocol following the implementation of a quality improvement intervention. The same criteria checklist was used to assess compliance across the preoperative, intraoperative, and postoperative phases. This phase aims to measure the impact of the training and identify improvements in compliance rates compared to the pre-intervention assessment.

INTERVENTIONS:
Other: ERAS Protocol Adaptation for Emergency Laparotomy — The intervention incorporated a comprehensive quality improvement approach, including a presentation, live demonstrations, and an instructional video to support the implementation of ERAS protocols. These methods emphasized the key components outlined by the ERAS ® Society guidelines for emergency laparotomy, ensuring that participants understood the importance of each protocol step and its application in clinical practice. As part of the quality improvement initiative, efforts were made to engage key stakeholders, including local governance and healthcare authorities, to align the intervention with policy frameworks. Training materials, including videos and manuals, were reviewed by a consultant surgeon to ensure accuracy and relevance. Additionally, a consultant surgeon conducted individual demonstrations in the operating room and ward, supplemented by weekly morning meetings with nurses, anesthesiologists, residents, and doctors for one month.
  Arms: Pre-Intervention Assessment of Staff Adherence to ERAS Protocol in Emergency Laparotomy

SUMMARY:
This study evaluates the implementation of Enhanced Recovery After Surgery (ERAS) protocols during emergency laparotomy procedures in a resource-limited hospital in Sudan. ERAS protocols are evidence-based guidelines designed to improve patient outcomes by reducing surgical stress and optimizing care across preoperative, intraoperative, and postoperative phases.

The audit will included adult patients and assessed adherence to ERAS society criteria tailored to local constraints. Data were collected through direct observations. A quality improvement and intervention was implemented, involving live demonstrations, instructional videos, and illustrated manuals to enhance staff understanding and compliance with the protocols.

By addressing gaps in protocol adherence and overcoming barriers such as resource limitations and knowledge gaps, the study highlights the feasibility of adapting ERAS protocols to emergency settings in low-resource environments, aiming to improve surgical care and patient outcomes.

DETAILED DESCRIPTION:
This study examines adherence to ERAS protocols during emergency laparotomy procedures in a resource-limited hospital in Sudan. While traditionally associated with elective surgeries, this study focuses on their adaptation to emergency laparotomies, which present unique challenges due to their urgency and complexity.

The study was conducted as a single-center, prospective clinical audit from, involving adult patients undergoing emergency laparotomy. The ERAS criteria assessed were tailored to the hospital's limited resources and encompassed criteria elements spanning preoperative, intraoperative, and postoperative phases. These criteria were designed to address critical aspects of patient care, such as early warning system usage, sepsis management, risk assessment, fluid and electrolyte correction, and patient education.

The study methodology included data collection in two phases: a pre-intervention phase to establish baseline compliance and a post-intervention phase following the implementation of a quality improvement initiative. The initiative involved extensive training for staff, including live demonstrations, instructional videos, and illustrated manuals, aimed at standardizing and improving protocol adherence.

Data collection was exclusively based on direct observation to assess adherence accurately while minimizing any observer effect that might alter staff behavior. Compliance with each criterion was assessed using a binary scoring system (compliant = 1, non-compliant = 0). The checklist was adapted from the ERAS Society guidelines, modified to fit the constraints of a low-resource setting, and underwent a pilot phase to ensure clarity and practicality.

The audit team consisted of eight members, including doctors, nurses, and an anesthesia technician, all trained to standardize data collection and scoring methods. Interventions emphasized practical applications of ERAS protocols in emergency settings and engaged key stakeholders to align improvements with institutional policies.

This study highlights the challenges of implementing ERAS protocols in resource-constrained environments, focusing on adapting these evidence-based practices to enhance patient care and improve surgical outcomes in emergency scenarios. By addressing barriers such as limited supplies, inadequate training, and workflow constraints, the study provides insights into the feasibility of scaling ERAS protocols in similar settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 59 years
* Underwent emergency laparotomy due to trauma

Exclusion Criteria:

* Patients who died during surgery or subsequent hospitalization
* Patients with incomplete medical records
* Patients who required re-laparotomy due to complications from previous surgeries
* Patients taking chronic anticoagulants

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The percentage of compliance with ERAS protocol criteria across preoperative, intraoperative, and postoperative phases. | From enrollment to 30 days post-intervention for each phase (pre-intervention and post-intervention phases)
  The percentage of compliance with ERAS protocol criteria across preoperative, intraoperative, and postoperative phases

CONTACTS AND LOCATIONS:
Overall Officials: Alsadig Suliman, MBBS, Msc, Principal Investigator — Sudan Medical Specialization Board; Aamir Hamza, Prof Surgery, Study Chair — University of Bahri
Locations (1):
- Alnao Teaching Hospital, Khartoum, Omdurman, Sudan

IPD SHARING:
Plan to Share IPD: No
Due to limitations in resources and infrastructure, we do not have a mechanism to securely share IPD at this time. Additionally, our ethical and regulatory approvals do not cover IPD sharing.